CLINICAL TRIAL: NCT05979675
Title: Acute Myeloid Leukemia Registry - Prospective National Multicentric Observational Study
Brief Title: Acute Myeloid Leukemia Registry
Acronym: AMLREGISTRY
Status: Recruiting | Type: Observational
Sponsor: Turkish Hematology Association (Other)
Responsible Party: Sponsor
Other Study IDs: AML_Registry
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All acute myeloid leukemia (AML) patients diagnosed after 1 Jan 2020 will be included to this study.

DETAILED DESCRIPTION:
This is a non interventional prospective disease registry, 250 prospective patients diagnosed with AML across 20 centers in Turkey.

Participating sites will consist of hematology clinics and routine follow-up procedures will be followed-up.

All patients diagnosed after 1 Jan 2020 as AML will be included and patients will be enrolled during 24 months of period and will be followed-up 36 months. Study will be completed in 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as AML after 1 Jan 2020
* Patients signed informed consent form

Exclusion Criteria:

* Patients under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All AML patients diagnosed after 1 Jan 2020 will be included to this study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2026-12-21 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 60 months
  From diagnosis to exits by any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Kurkcu, Study Director — Sentez Cro
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakus V, Pinar IE, Iltar U, Yenihayat EM, Polat MG, Celik S, Malkan UY, Cengiz Seval G, Dogan A, Akdeniz A, Ozbalci D, Ince I, Erdem R, Mehtap O, Kirkizlar HO, Kacmaz M, Deveci B, Aykas F, Korkmaz G, Yigit Kaya S, Afacan Ozturk HB, Sevindik OG, Can F, Cekdemir D, Aslan C, Bulbul H, Karabulut ZT, Maral S, Durusoy SS, Demirkan F, Goker H, Ozkalemkas F, Keklik M, Toprak SK, Karatas AF, Atas U, Alacacioglu I; Turkish Society of Hematology-Acute Leukemias Working Group. Clinical Characteristics, Treatment Approaches, and Survival Predictors in Adult Acute Myeloid Leukemia: Interim Results from the Turkish Society of Hematology AML Registry. J Clin Med. 2025 Oct 18;14(20):7367. doi: 10.3390/jcm14207367. PMID 41156238
- [Derived] Pinar IE, Celik S, Polat MG, Karatas AF, Dogan A, Iltar U, Cengiz Seval G, Malkan UY, Ince I, Yenihayat EM, Akdeniz A, Kacmaz M, Erdem R, Afacan Ozturk HB, Kirkizlar HO, Korkmaz G, Aykas F, Mehtap O, Deveci B, Sevindik OG, Can F, Ozbalci D, Bulbul H, Durusoy SS, Atas U, Keklik M, Toprak SK, Goker H, Demirkan F, Ozkalemkas F, Alacacioglu I, Karakus V; Turkish Society of Hematology-Acute Leukemias Working Group. Comprehensive analysis of FLT3-mutated patients with acute myeloid leukemia with updated 2022 European LeukemiaNet recommendations: insights from the Turkish AML registry project. BMC Cancer. 2025 Oct 10;25(1):1546. doi: 10.1186/s12885-025-14987-z. PMID 41073967